CLINICAL TRIAL: NCT03139123
Title: Prevalence of Hypotension Associated With Preload Dependence During Continuous Renal Replacement Therapy
Acronym: PRELOAD-CRRT
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL17_0120
Record Dates: First submitted 2017-04-27; First posted 2017-05-03 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Kidney Injury; Renal Failure, Acute
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with acute kidney injury: Intensive care unit patients with acute kidney injury. Patients under continuous renal replacement therapy and hemodynamic monitoring.
  Interventions: Other: Hemodynamic monitoring during passive leg raising

INTERVENTIONS:
Other: Hemodynamic monitoring during passive leg raising — Measurement of hypotensive episodes related to preload dependance.

SUMMARY:
Per-dialytic hypotension is common in Intensive Care Unit patients under continuous renal replacement therapy, and occurs in nearly 50% of the patients. To date, there is a lack of study having characterized the underlying mechanism of hypotension in this setting. New diagnostic methods are now available with high reliability to identify hypovolemia as the underlying cause of hypotension, among which change in cardiac index during passive leg raising may be the less affected by restrictive validity criteria. A change in cardiac index greater than 10% during this test is highly predictive of preload dependence, i.e the probability than cardiac index will increase if cardiac preload increases.

The aim of this study is then to identify, among hypotensive episodes occurring during renal replacement therapy in Intensive Care Unit patients, the percentage of episodes related to preload dependence as identified by passive leg raising.

ELIGIBILITY:
Inclusion Criteria:

* Intensive Care Unit patients with acute kidney injury
* under continuous renal replacement therapy initiated since less than 24 hours
* under hemodynamic monitoring by the PiCCO® device.

Exclusion Criteria:

* lower limb amputation
* inferior vena cava compression
* intracranial hypertension
* age below 18 year
* pregnancy
* advance directives to withhold or withdraw life sustaining treatment,
* lack of written informed consent by patient or next of kin
* lack of affiliation to social security as required by French regulation
* patient under a legal protective measure
* previous inclusion in current study
* inclusion in another research study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study concerns patients hospitalized in intensive care unit at the Croix-Rousse hospital in Lyon with acute renal insufficiency (stage 3 of the Kidney Disease: Improving Global Outcomes classification) for which treatment with continuous hemofiltration was initiated less than 24 hours ago and for whom a hemodynamic monitoring device (PiCCO® device) has been implanted due to acute circulatory failure and is functional.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2017-05-18 (Actual); Primary Completion 2020-08-29 (Actual); Study Completion 2020-11-21 (Actual)

PRIMARY OUTCOMES:
Presence of hypotensive episode by hemodynamic monitoring | 7 days
  An hypotensive episode is defined as mean arterial pressure < 65 mm Hg and one of the following events :
  * Fluid administration
  * OR increase of vasopressor dose
  * OR decrease of fluid removal
Preload dependence identified by cardiac index greater than 10% during passive leg raising | 7 days
  The passive leg raising allows to identify the percentage of hypotensive episodes related to preload dependence.
  A change in cardiac index greater than 10% during this test is highly predictive of preload dependence, i.e the probability than cardiac index will increase if cardiac preload increases.

CONTACTS AND LOCATIONS:
Locations (1):
- Service de réanimation médicale- Hôpital de la Croix-Rousse, Lyon, France

REFERENCES:
- [Derived] Bitker L, Biscarrat C, Yonis H, Chivot M, Chauvelot L, Chazot G, Mezidi M, Deniel G, Richard JC. Determinants of Urine Output Using Advanced Hemodynamic Monitoring in Critically Ill Patients Undergoing Continuous Renal Replacement Therapy. Blood Purif. 2024;53(3):189-199. doi: 10.1159/000535544. Epub 2023 Dec 16. PMID 38104538